CLINICAL TRIAL: NCT00274508
Title: Effect of Tiotropium on Exercise Tolerance and Static and Dynamic Lung Volumes in COPD Patients (A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study)
Brief Title: Effect of Tiotropium (Spiriva) on Exercise Tolerance in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.223
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium bromide

SUMMARY:
To investigate whether tiotropium (Spiriva) improves exercise endurance in patients with COPD

ELIGIBILITY:
Inclusion criteria:

Male or female patients with a clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD) based on American Thoracic Society (ATS) guidelines with:

* Relatively stable, moderate to severe airway obstruction with an Forced Expiratory Volume in One Second (FEV1) less than or equal to 65% of predicted normal (determined at Visit 1).
* Presence of lung hyperinflation as demonstrated by Functional Residual Capacity determined by body plethysmography (TGV(FRC)) greater than or equal to 120% of predicted normal (determined at Visit 1).
* Age greater or equal to 40 years and less than or equal to 75 years.
* A cigarette smoking history of more than ten pack-years. A pack-year was defined as the equivalent of smoking one pack of cigarettes per day for a year.
* Able to perform all specified procedures and able to maintain all necessary records during the study period as required in the protocol.
* Able to inhale the trial medication from the HandiHaler device.

Exclusion criteria:

* Patients with a significant disease other than COPD. A significant disease was defined as a disease which, in the opinion of the investigator, may have put the patient at risk because of participation in the trial or may have influenced the results of the trial or the patient's ability to participate in the trial.
* Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defined a disease listed as an exclusion criterion, the patient was excluded.
* Patients with Serum Glutamic Oxaloacetic Transaminase (SGOT) ≥1.5 x ULN (upper limit of normal range), Serum Glutamic Pyruvic Transaminase (SGPT) ≥1.5 x ULN bilirubin ≥1.5 x ULN or creatinine ≥1.5 x ULN were excluded regardless of the clinical condition.
* Patients with a recent history (i.e., 1 year or less) of myocardial infarction.
* Patients with a recent history (i.e., 3 years or less) of heart failure, pulmonary edema, or patients with cardiac arrhythmia (with or without symptoms) or any contraindication to exercise.
* Patients requiring the regular use of daytime oxygen therapy.
* Patients with known active tuberculosis.
* Patients with a history of cancer within the last 5 years. Patients with treated basal cell carcinoma were eligible.
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
* Patients who had undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons were evaluated as per the first exclusion criterion (i.e., significant disease other than COPD).
* Patients with an upper respiratory tract infection in the 6 weeks prior to the Screening Visit (Visit 1) or during the run-in period.
* Further exclusion criteria apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2000-10-10 (Actual); Primary Completion 2003-01-07 (Actual)

PRIMARY OUTCOMES:
Endurance time during a constant work rate exercise test to symptom limitation | 2 hours and 15 minutes after trial medication administration on Day 42

SECONDARY OUTCOMES:
Constant work rate exercise test to symptom limitation | 8 hours post-dose after 6 weeks of treatment
Breathing discomfort during constant work rate exercise test as measured by the modified Borg Scale | 6 weeks
Dynamic lung hyperinflation during exercise as determined by IRVdyn (IC minus VT) and EELVdyn (TLC) | 6 weeks
Evaluation of VE and VEcap during exercise (selected centers) | 6 weeks
Evaluation of static lung hyperinflation as measured by RV/TLC and by TGV(FRC)/TLC | 6 weeks
Evaluation of TAC (TAV = TLC(BOX)-VA(IG)) | 6 weeks
Evaluation of slow vital capacity (SVC) | 6 weeks
Evaluation of maximal expiratory flow rates and volumes FEV1, FVC, FEF25-75%, FEF50%, FEF75%, SVC | 6 weeks
Evaluation of TGV, Raw, SGaw and RV | 6 weeks
Evaluation of SaO2, VO2, VCO2, Ti, Te, VE, VT, breathing frequency (f) during constant work rate exercise test | 6 weeks
Physician's Global Assessment | 6 weeks
Assessement of Pulse/heart rate and blood pressure in conjunction with spirometry and exercise | 6 weeks
Changes in Physical examination and ECG | 6 weeks
Occurrence of Adverse Events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (28):
- United States (4):
  - St. Elizabeth's Medical Center of Boston, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - St. Thomas Health Services, Nashville, Tennessee
  - Presbyterian Hospital of Dallas, Dallas, Texas
- Australia (5):
  - Phase I Unit, Randwick, New South Wales
  - Immunology Department, Westmead, New South Wales
  - Department of Respiratory Medicine, Daw Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Department of Respiratory Medicine, Heidelberg, Victoria
- Canada (13):
  - Respiratory Research, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Respiratory Clinic, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - Cardio Repiratory, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - 1053 Carling Avenue, Ottawa, Ontario
  - Department of Respiratory Medicine, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Montreal Chest Institute - McGill University Health Centre, Montreal, Quebec
  - Pulmonary Function Lab, Montreal, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Germany (6):
  - Klinikum der Universität zu Köln, Cologne
  - Pneumologisches Forschungsinstitut GmbH am Krankenhaus, Hamburg
  - Fraunhofer-Institut für Toxikologie und, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Neurologische Klinik der Otto-von-Guericke-Universität, Magdeburg
  - Boehringer Ingelheim Investigational Site, München